CLINICAL TRIAL: NCT02047058
Title: A Multi-center, Prospective, Observational Study of Analysis of Q Cell Markers in Patients With Newly Diagnosed Primary Glioblastoma (Phase IV)
Brief Title: Treatment Response and Prognosis in Glioma Patients: Q Cell and Its Biological Characteristics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou General Hospital of Guangzhou Military Command (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Capital Medical University (Other); Tianjin Medical University General Hospital (Other); Shenzhen Second People's Hospital (Other); Huashan Hospital (Other); West China Hospital (Other); Xiangya Hospital of Central South University (Other); The First Hospital of Jilin University (Other); First Hospital of China Medical University (Other); Qilu Hospital of Shandong University (Other); Second Affiliated Hospital of Soochow University (Other); Sun Yat-sen University (Other); Guangzhou First People's Hospital (Other); Xi'an Jiaotong University (Other); Southern Medical University, China (Other); Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFGC-001-MCP
Record Dates: First submitted 2014-01-21; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Glioblastoma; Malignant Glioma
Keywords: biomarker; Q cell; Overall survival; Progression-free survival
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — tumor sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- high-risk: high-risk is determined by the evaluation of the biomarkers of Q cell.

SUMMARY:
The purpose of this study is to determine whether Q cells separated from the glioma sample are determinants in treatment response and prognosis of glioma patients

DETAILED DESCRIPTION:
The unique markers of Qcell were screened using the method of genomics and

proteomics, then these markers will be qualitatively and quantitatively evaluated in

glioblastoma patients by comparing their relationship with overrall

survival/progression-free survival and treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. >=18 years old
2. Primary Glioblastoma is newly diagnosed and confirmed histologically
3. Patient is expected to be treated with temozolomide and followed up routinely at the study site.
4. Willing to sign the informed consent

Exclusion Criteria:

1. Currently enrolled in any other clinical study
2. History of any other malignancies
3. Refusal to give consent
4. No available tumor tissue for IDH analysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with glioblastoma undergo operation and sufficient tumor specimens
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The effect of each single molecular marker of Q cell on progression-free survival | 3-5 days postoperatively
  Participating centres collected data and submitted it by Email to the coordinating centre at the Nanfang Glioma Center. 300 patients with glioblastoma will be prospectively enrolled in this study. The unique markers of Q cell which had been screened using the method of genomics and proteomics will be measured and compared with progression-free and overall survival of patients. Regrettably,the markers of Q cell cannot yet be disclosed because of the confidentiality requirement. Progression-free survival (PFS) will be calculated from the day of ﬁrst surgery until tumor progression, death, or end of follow-up. Overall survival (OS) will be calculated from the day of ﬁrst surgery until death or end of follow-up. The effect of each single molecular marker on PFS and OS was investigated using the Cox proportional hazards model.
The effect of each single molecular marker of Q cell on overall survival | 3-5 days postoperatively
  Participating centres collected data and submitted it by Email to the coordinating centre at the Nanfang Glioma Center. 300 patients with glioblastoma will be prospectively enrolled in this study. The unique markers of Q cell which had been screened using the method of genomics and proteomics will be measured and compared with progression-free and overall survival of patients. Regrettably,the markers of Q cell cannot yet be disclosed because of the confidentiality requirement. Progression-free survival (PFS) will be calculated from the day of ﬁrst surgery until tumor progression, death, or end of follow-up. Overall survival (OS) will be calculated from the day of ﬁrst surgery until death or end of follow-up. The effect of each single molecular marker on PFS and OS was investigated using the Cox proportional hazards model.

SECONDARY OUTCOMES:
We will correlate molecular markers of Q cell with other genetic alterations | 3-5 days postoperatively
  Other genetic alterations which have been previously reported include isocitrate dehydrogenase mutation, o6-methylguanine-DNA-methyltransferase methylation, 1p19q co-delation, Tumor Protein 53 (TP53) mutation, histone H3.3 (H3F3A) mutations, etc. The Chi-square test will be used to compare the genotype distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Songtao Qi, Doctor, Principal Investigator — Nanfang Glioma centre, Guangzhou, China
Locations (1):
- Nanfang Glioma Centre, Guangzhou, Guangdong, China

REFERENCES:
- [Background] SongTao Q, Lei Y, Si G, YanQing D, HuiXia H, XueLin Z, LanXiao W, Fei Y. IDH mutations predict longer survival and response to temozolomide in secondary glioblastoma. Cancer Sci. 2012 Feb;103(2):269-73. doi: 10.1111/j.1349-7006.2011.02134.x. Epub 2011 Nov 28. PMID 22034964
- [Background] Qi ST, Yu L, Lu YT, Ou YH, Li ZY, Wu LX, Yao F. IDH mutations occur frequently in Chinese glioma patients and predict longer survival but not response to concomitant chemoradiotherapy in anaplastic gliomas. Oncol Rep. 2011 Dec;26(6):1479-85. doi: 10.3892/or.2011.1428. Epub 2011 Aug 19. PMID 21874255
- [Background] Sturm D, Witt H, Hovestadt V, Khuong-Quang DA, Jones DT, Konermann C, Pfaff E, Tonjes M, Sill M, Bender S, Kool M, Zapatka M, Becker N, Zucknick M, Hielscher T, Liu XY, Fontebasso AM, Ryzhova M, Albrecht S, Jacob K, Wolter M, Ebinger M, Schuhmann MU, van Meter T, Fruhwald MC, Hauch H, Pekrun A, Radlwimmer B, Niehues T, von Komorowski G, Durken M, Kulozik AE, Madden J, Donson A, Foreman NK, Drissi R, Fouladi M, Scheurlen W, von Deimling A, Monoranu C, Roggendorf W, Herold-Mende C, Unterberg A, Kramm CM, Felsberg J, Hartmann C, Wiestler B, Wick W, Milde T, Witt O, Lindroth AM, Schwartzentruber J, Faury D, Fleming A, Zakrzewska M, Liberski PP, Zakrzewski K, Hauser P, Garami M, Klekner A, Bognar L, Morrissy S, Cavalli F, Taylor MD, van Sluis P, Koster J, Versteeg R, Volckmann R, Mikkelsen T, Aldape K, Reifenberger G, Collins VP, Majewski J, Korshunov A, Lichter P, Plass C, Jabado N, Pfister SM. Hotspot mutations in H3F3A and IDH1 define distinct epigenetic and biological subgroups of glioblastoma. Cancer Cell. 2012 Oct 16;22(4):425-37. doi: 10.1016/j.ccr.2012.08.024. PMID 23079654